CLINICAL TRIAL: NCT07272057
Title: The Impact of SGLT2i on the Outcome of Advanced Lung Cancer in Patients With Diabetes
Brief Title: SGLT2 Inhibitors and Survival in Lung Cancer Patients With Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Liang Zhao, Dr, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLC-DO
Record Dates: First submitted 2025-11-18; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Sodium-Glucose Transporter 2 Inhibitors; salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): On the basis of standard cancer treatment, take dapagliflozin for at least three months, once a day, 10 mg each time.
  Interventions: Drug: SGLT-2 inhibitor
- control group (Sham Comparator): Based on the standard treatment for tumors, for the treatment of diabetes, no dapagliflozin has been taken.
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Drug: SGLT-2 inhibitor — SGLT2 inhibitors used for patients with lung cancer and diabetes
  Arms: treatment group
Other: Sham (No Treatment) — SGLT2 inhibitors are not used for patients with lung cancer and diabetes
  Arms: control group

SUMMARY:
The goal of this clinical trial

The goal of this clinical trial is to evaluate whether SGLT2 inhibitor drugs can extend overall survival or delay the progression of the tumor in patients with both advanced lung cancer and diabetes. It will also check if these drugs are safe for these patients. The main questions it aims to answer are:

* Does adding an SGLT2 inhibitor to standard cancer treatment improve survival?
* Does it cause more or fewer cardiovascular toxicity?
* What side effects do participants experience? Researchers will compare a group taking an SGLT2 inhibitor to a group not taking SGLT2 inhibitor to see if the drug works.

Participants will:

* Be adults diagnosed with advanced lung cancer and type 2 diabetes.
* Take either the SGLT2 inhibitor pill or other hypoglycemic drugs once a day alongside their cancer treatment.
* Undergo regular clinical visits for monitoring, laboratory tests, and imaging studies

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer patients receiving standard anti-tumor treatment; type 2 diabetes; patients with a score of 0-2 assessed by Eastern Cooperative Oncology Group's performance status; the patients agreed to participate in this study.

Exclusion Criteria:

* Severe abnormalities in liver, kidney or heart functions; expected lifespan less than 3 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-07 (Estimated); Primary Completion 2026-10-07 (Estimated); Study Completion 2026-11-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with death | From enrollment to the end of treatment at 12 months

SECONDARY OUTCOMES:
Number of Participants with new-onset atrial fibrillation/flutter, acute coronary syndrome, myocarditis, massive pericardial effusion, heart failure and third-degree atrioventricular block. | From enrollment to the end of treatment at 12 months

IPD SHARING:
Plan to Share IPD: No